CLINICAL TRIAL: NCT01815489
Title: Molecular Analysis of Microbial DNA in Infected Necrotizing Pancreatitis
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: California HealthCare Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CHS-001
Record Dates: First submitted 2012-08-01; First posted 2013-03-21 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2014-05

CONDITIONS: Necrotizing Pancreatitis
Keywords: Necrotizing Pancreatitis; Pancreatitis; Infection; Bacteria; Microbiology
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Pancreatitis; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripancreatic fluid, pancreatic tissue, blood sample, stool sample
Oversight: Data Monitoring Committee: No

SUMMARY:
Necrotizing pancreatitis is a severe form of inflammation of the pancreas with subsequent destruction of the pancreas (necrosis). Often, this condition manifests in patients as an overwhelming systemic inflammatory response and multisystem organ failure. Many times the pancreas can become superinfected with bacteria and other organisms as a result of this process. Clinicians may decide to sample fluid from the pancreas or pancreatic tissue to determine the presence of infection. This can be done through surgery with a concurrent debridement and drainage of the pancreas or by a radiologist using an ultrasound or CT guided method to sample the pancreatic fluid. These samples are then sent for culture in the microbiology laboratory. Culture results often reveal 1-2 types of infecting bacteria that originate from the gastrointestinal tract. The investigators hypothesize that in actuality, many different kinds of bacteria may infect the pancreas. This project uses molecular DNA techniques to help identify bacteria present in the pancreas of patients with severe necrotizing pancreatitis.

DETAILED DESCRIPTION:
In this study, patients with severe necrotizing pancreatitis will be followed prospectively throughout their hospital course (anticipated duration of hospitalization ranging between 4-8 weeks). If patients are suspected to have infection of pancreatic necrosis, they will be consented for enrollment. Patients will be determined by their attending physician to require either operative intervention or radiologic guided drainage of pancreatic necrosis and infected peripancreatic fluid. At the time of drainage procedure or intervention, one sample of peripancreatic fluid will be sent to the hospital's microbiology department for standard gram stain and bacterial culture identification and a second sample will be frozen for bacterial DNA analysis. Patients will be followed for the duration of their hospitalization for in hospital outcomes, mortality and final microbiology culture results. Samples will then be processed at six months and one year following sample collection for bacterial DNA deep sequencing analysis and will be compared to bacteria identified using standard culture technique.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Severe necrotizing pancreatitis as evidenced by clinical examination, biochemical analysis, and/or imaging studies demonstrating pancreatitis and pancreatic necrosis

Exclusion Criteria:

* Age less than 18 years old
* Participation in another device or drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults over 18 years of age with a diagnosis of necrotizing pancreatitis and concern for superinfection of the pancreas related to their condition.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Bacteria | June 2012
  Bacteria present in peri-pancreatic fluid and pancreatic tissue will be analyzed and identified suing molecular based methods. Comparisons will be made to bacteria identified using standard culture techniques.

SECONDARY OUTCOMES:
Cytokines | June 2012
  Blood samples will be taken from each patient to measure the level of different cytokines at the time of sample collection
Gastrointestinal Bacterial Flora | June 2012
  A small stool sample will be taken from each patient to determine normal GI flora that may be translocating to the pancreas in patients with severe pancreatitis.

CONTACTS AND LOCATIONS:
Overall Officials: David Iannitti, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States